CLINICAL TRIAL: NCT06491303
Title: Study of Effects of Levetiracetam Monotherapy on Various Hematological Parameters in Adult Patients Suffering of Epilepsy
Brief Title: Effects of Levetiracetam Monotherapy on Various Hematological Parameters in Adult Patients Suffering of Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa AA Khaled, professor, Assiut University
Other Study IDs: Levetiracetam
Record Dates: First submitted 2024-05-20; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Neutropenia; Thrombocytopenia; Aplastic Anemia; Anemia; Epilepsy
Keywords: Levetiracetam; Hematological effects; antiepileptic drugs; Epilepsy; Neutropenia; Thrombocytopenia
MeSH Terms: conditions — Neutropenia; Thrombocytopenia; Anemia, Aplastic; Anemia; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Distribution of studied patients by age in years.: Adult patients suffering of epilepsy aged 18 to 60 years old
- Distribution of studied patients by duration of levetiracetam administration in months: Adult patients suffering of epilepsy and receiving treatment of levetiracetam for at least 6 months

SUMMARY:
Low therapeutic index of established antiepileptic drugs (AEDs) coupled with better understanding of the pathophysiology of seizure has encouraged the development of several novel AEDs. The conventional antiepileptics like phenytoin, phenobarbitone, valproate and carbamazepine and newer antiepileptics like levetiracetam. are used for epilepsy. AEDs induce potentially toxic effects over a period of time which remains undetermined over very long time. Earlier studies in this regard, states uneven results about hematological (Hb%, blood cell count etc.) toxicity of AEDs.

DETAILED DESCRIPTION:
Epilepsy is a chronic neurologic disease that is considered the most common neurological diseases in the world and comes third after cerebrovascular and Alzheimer's disease. Epilepsy is a disorder characterized by a long-term tendency to cause epileptic seizures due to abnormal electrical activity in the brain with neurological, cognitive, psychological and social consequences . However, it is not a single disease entity but it is a collection of different kinds of seizures resulting from several mechanisms and different cause. The aim of epilepsy management is complete seizures cessation and maintenance of a good quality of life, which is affected not only by the epileptic attacks but also by the adverse effect of the drugs used .Levetiracetam (LEV) is a relatively new, broad-spectrum AED that has seen extensive use during recent years . Its mechanism of action is not completely known, but differs from those of other AEDs. LEV is described as being well tolerated, and the most common adverse effects are generally mild . Studies evaluating the effect of levetiracetam on hematological parameters have reported a spectrum of hematological abnormalities that ranges from mild thrombocytopenia or neutropenia to anemia, red cell aplasia, until bone marrow failure. Fortunately, potentially fatal hematological disorders such as aplastic anemia are very rare.

ELIGIBILITY:
Inclusion Criteria: Adult Epileptic patients of both genders aged >18 years on mono-therapy of levetiracetam anti-epileptic drug treatment for at least six months.

Exclusion Criteria:

1. Patients were on treatment for less than six months.
2. Patients had other conditions besides epilepsy that could affect blood parameters.
3. patients on treatment with other antiepileptic medications besides levetiracetam.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Based on determining the main outcome variable, The estimated minimum required sample size is 45 patients. The sample size was calculated using Epi-info version 7 software, based on the following assumptions: Main outcome variable is to investigate hematological changes in adult patients with epilepsy who were treated with levetiracetam as monotherapy. Based on previous studies [8] the percentage of patients who their hemoglobin fell below 10g/dl while taking Levetiracetam was 8%, and based on the percentage confidence limits of 5% and a Confidence level=80%
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Study of Effects of Levetiracetam Monotherapy on Various Hematological Parameters in Adult Patients Suffering of Epilepsy | one years
  All 45 patients will be included within certain inclusion criteria after informed consent will be subjected to full history, general examination,systemic examination including cardiac, chest and abdominal examination will be done to detect associated or excluded conditions and Laboratory tests include complete blood count assay.
  The primary outcome measures to be assessed in this study is the effect of Levetiracetam(at least 6 months duration of treatment)on complete blood count including
  1. Haemoglobin level.
  2. Red cell count.
  3. Hematocrit value.
  4. M.C.V
  5. M.C.H
  6. M.C.H.C
  7. Platelets count including MPV and PCT.
  8. Total leucocytic count including neutrophils(band and segmented), lymphocytes, monocytes, basophils and eosinophils.

CONTACTS AND LOCATIONS:
Overall Officials: Safa Abdel-Sattar, professor, Study Director — Assiut University; Rania Mohamed, professor, Study Director — Assiut University

REFERENCES:
- [Background] Attilakos A, Dinopoulos A, Paschalidou M, Tsirouda M, Karalexi M, Prasouli A, Garoufi A. Long-term effect of levetiracetam monotherapy on haematological parameters in children with epilepsy: A prospective study. Epilepsy Res. 2018 Sep;145:160-162. doi: 10.1016/j.eplepsyres.2018.07.001. Epub 2018 Jul 6. PMID 30007241
- [Background] Dinopoulos A, Attilakos A, Paschalidou M, Tsirouda M, Garoufi A, Moustaki M, Siafakas N, Papaevangelou V. Short-term effect of levetiracetam monotherapy on haematological parameters in children with epilepsy: a prospective study. Epilepsy Res. 2014 May;108(4):820-3. doi: 10.1016/j.eplepsyres.2014.02.006. Epub 2014 Feb 19. PMID 24630047